CLINICAL TRIAL: NCT00425854
Title: An Open Label Phase II Trial to Assess the Efficacy and Safety of a Once Daily Oral Dose of 50 mg BIBW 2992 in Two Cohorts of Patients With HER2-negative Metastatic Breast Cancer After Failure of no More Than Two Chemotherapy Regimen
Brief Title: An Open Label Phase II Trial of BIBW 2992 in Patients With HER2-negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1200.10; 2006-002018-36 (EudraCT Number: EudraCT)
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-08

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Afatinib

ARMS (1):
- BIBW 2992 (Experimental): high dose once daily
  Interventions: Drug: BIBW 2992

INTERVENTIONS:
Drug: BIBW 2992 — high dose once daily

SUMMARY:
The purpose of this trial is to evaluate the efficacy, safety and pharmacokinetics of BIBW 2992, a dual, irreversible EGFR- and HER2-inhibitor, in two cohorts of patients with HER2-negative breast cancer after failure of no more than three regimen of prior chemotherapy.

ELIGIBILITY:
Inclusion criteria:

Inclusion Criteria:

* Female patients age 18 years or older
* Histologically proven breast cancer after failure or relapse of no more than three lines of chemotherapy including adjuvant, irrespective of prior hormone therapy metastatic disease (stage IV);
* HER2-negative patients (HER2 1+ or negative, or HER2 2+ and FISH negative)
* At least one measurable tumour lesion (RECIST);
* Availability of tumour samples
* Written informed consent that is consistent with ICH-GCP guidelines and local law
* Eastern Cooperative Oncology Group (ECOG, R01-0787) performance score 0 - 2.

Exclusion criteria:

Exclusion Criteria:

* Active infectious disease
* Gastrointestinal disorders that may interfere with the absorption of the study drug or chronic diarrhoea
* Serious illness, concomitant non-oncological disease or mental problems considered by the investigator to be incompatible with the protocol
* Active/symptomatic brain metastases
* Cardiac left ventricular function with resting ejection fraction < 50% (below upper limit of normal)
* ANC less than 1500/mm3 platelet count less than 100 000/mm3
* Bilirubin greater than 1.5 mg /dl (>26 and#61549 mol /L, SI unit equivalent)
* AST and ALT greater than 2.5 times the upper limit of normal or greater 5 times the upper limit of normal in case of known liver metastases
* Serum creatinine greater than 1.5 mg/dl (>132 and#61549 mol/L, SI unit equivalent)
* Patients who are sexually active and unwilling to use a medically acceptable method of contraception
* Pregnancy or breast-feeding
* Concomitant treatment with other investigational drugs or other anti-cancer-therapy during this study and/or during the past two/four weeks, prior to the first treatment with the trial drug. Concurrent treatment with biphosphonates is allowed
* Previous treatment with trastuzumab, EGFR-, or EGFR/HER2-inhibitors patients unable to comply with the protocol
* Active alcohol or drug abuse
* Other malignancy within the past 5 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-11; Primary Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (14):
- Belgium (6):
  - 1200.10.3201 Boehringer Ingelheim Investigational Site, Brussels
  - 1200.10.3208 Boehringer Ingelheim Investigational Site, Brussels
  - 1200.10.3203 Boehringer Ingelheim Investigational Site, Charleroi
  - 1200.10.3205 Boehringer Ingelheim Investigational Site, Ghent
  - 1200.10.3204 Boehringer Ingelheim Investigational Site, Leuven
  - 1200.10.3206 Boehringer Ingelheim Investigational Site, Wilrijk
- Germany (8):
  - 1200.10.49005 Boehringer Ingelheim Investigational Site, Berlin
  - 1200.10.49007 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1200.10.49008 Boehringer Ingelheim Investigational Site, Erlangen
  - 1200.10.49010 Boehringer Ingelheim Investigational Site, Essen
  - 1200.10.49003 Boehringer Ingelheim Investigational Site, Kiel
  - 1200.10.49004 Boehringer Ingelheim Investigational Site, Mainz
  - 1200.10.49001 Boehringer Ingelheim Investigational Site, München
  - 1200.10.49006 Boehringer Ingelheim Investigational Site, Wiesbaden

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Patients with human epidermal growth factor 2- (HER2-) negative, oestrogen receptor- (ER-) negative, progesterone- (PgR-) negative tumours (triple negative tumours) receiving oral dose of Afatinib 50 mg once daily (qd)
- Cohort B: Patients with HER2-negative, ER-positive and/or PgR-positive tumours receiving oral dose of Afatinib 50 mg qd
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 29 (Treated) | 21 (Treated)
Completed | 0 (On treatment at analysis cut-off date (30 Sep 2009)) | 0 (On treatment at analysis cut-off date (30 Sep 2009))
Not Completed | 29 | 21
Not completed — Progressive Disease | 19 | 12
Not completed — Dose reduction toxicity AE | 8 | 7
Not completed — Other Adverse Event | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 29 | 21 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (11.5) | 61.0 (14.3) | 57.1 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 21 | 50
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Clinical Benefit (CB)
Description: CB was defined as CR, PR or stable disease (SD) for a minimum of 4 months (modified CB) and was assessed according to RECIST 1.0 criteria. CB was secondary endpoint only for Cohort B as it was primary endpoint for Cohort A.
Time Frame: Tumour assessments were performed at screening, week 8, week 16, week 24, and every 8 weeks thereafter.
Description (as registered): CB was defined as CR, PR or stable disease (SD) for a minimum of 4 months (modified CB) and was assessed according to RECIST 1.0 criteria. CB was primary endpoint only for Cohort A.
Population: TS. No data for Cohort A as CB was secondary endpoint only for Cohort B.
Measure: Number; unit: Participants with CB
Arm/Group | Cohort B
Number analyzed (Participants) | 21
Participants with CB
  With CB | 1
  Without CB | 17
  missing | 3
Statistical Analysis 1: Comparison: Cohort B; Test type: Superiority or Other; Maximum Likelihood = 0.048, 95% CI 2-sided [0.001 to 0.238] — Maximum Likelihood estimates. The clinical benefit rate for Cohort A was calculated by relating the number of patients with CB to all treated patients in Cohort B. The CI is an exact Clopper Pearson CI

2. Secondary Outcome: Time to OR
Description: The time to OR was the duration from the first treatment to the time when the measurement criteria for CR and/or PR were met according to RECIST 1.0 criteria.
Time Frame: Tumour assessments were performed at screening, week 8, week 16, week 24, and every 8 weeks thereafter.
Population: TS. Median time to OR was not calcuable as there was no OR observed.
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Duration of OR
Description: Duration of OR was measured from the time the criteria for CR or PR (whichever was documented first) were first met until the first date that progressive disease or death was objectively documented.
Time Frame: Tumour assessments were performed at screening, week 8, week 16, week 24, and every 8 weeks thereafter.
Population: TS. Median duration of OR was not calcuable as there was no OR observed.
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the first treatment to the occurrence of tumour progression or death, whichever came first. It was assessed according to RECIST 1.0 criteria as well as by the investigators assessment. Median time results from unstratified Kaplan-Meier estimates.
Time Frame: Tumour assessments were performed at screening, week 8, week 16, week 24, and every 8 weeks thereafter.
Population: TS
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 29 | 21
days | 52 [39 to 71] | 54 [50 to 112]

5. Primary Outcome: Objective Response (OR)
Description: OR is defined as complete response (CR) and partial response (PR) and was assessed according to the Response Evaluation Criteria in Solid Tumours version 1.0 (RECIST). OR was primary endpoint only for Cohort B.
Time Frame: Tumour assessments were performed at screening, week 8, week 16, week 24, and every 8 weeks thereafter.
Population: Treated Set (TS). TS consisted of all patients who received at least one dose of trial medication. No data for Cohort A as OR was primary endpoint only for Cohort B.
Measure: Number; unit: Participants with OR
Arm/Group | Cohort B
Number analyzed (Participants) | 21
Participants with OR | 0

6. Primary Outcome: Clinical Benefit (CB)
Description: CB was defined as CR, PR or stable disease (SD) for a minimum of 4 months (modified CB) and was assessed according to RECIST 1.0 criteria. CB was primary endpoint only for Cohort A.
Time Frame: Tumour assessments were performed at screening, week 8, week 16, week 24, and every 8 weeks thereafter.
Description (as registered): CB was defined as CR, PR or stable disease (SD) for a minimum of 4 months (modified CB) and was assessed according to RECIST 1.0 criteria. CB was secondary endpoint only for Cohort B as it was primary endpoint for Cohort A.
Population: TS. No data for Cohort B as CB was primary endpoint only for Cohort A.
Measure: Number; unit: Participants
Arm/Group | Cohort A
Number analyzed (Participants) | 29
Participants
  With CB | 3
  Without CB | 24
  missing | 2
Statistical Analysis 1: Comparison: Cohort A; Test type: Superiority or Other; Maxium Likelihood; Clinical benefit rate = 0.10, 95% CI 2-sided [0.02 to 0.27] — Maximum Likelihood estimates. The clinical benefit rate for Cohort A was calculated by relating the number of patients with CB to all treated patients in Cohort A. The confidence interval (CI) is an exact Clopper Pearson CI

7. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from randomisation to death.
Time Frame: From randomisation to end of follow-up.
Population: TS. As only 9 patient (31 percent) of Cohort A had died the median OS time was not estimable for Cohort A.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 29 | 21
days | NA [120 to NA] — The 95% confidence interval is actually 120 to infinity, a median is not available. | 448 [310 to 537]

8. Secondary Outcome: Significant Change in Cardiac Left Ventricular Ejection Fraction (LVEF)
Description: LVEF as measured by echocardiography or Multiple Gated Acquisition (MUGA) scan. MUGA scan is an useful noninvasive tool for assessing the function of the heart. Significant change in LVEF values was defined as >=20 percent decrease from baseline or to below lower limit of normal, which was defined as 50 percent.
Time Frame: Baseline and last assessment
Population: TS
Measure: Number; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 29 | 21
Participants | 1 | 2

9. Secondary Outcome: Best Change From Baseline in ECOG Performance Status
Description: Best change from baseline in ECOG (Eastern Cooperative Oncology Group) performance status. ECOG is measured as score between 0 (fully active) and 5 (dead).
Time Frame: baseline till end of treatment
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 29 | 21
participants
  improved | 1 | 0
  deteriorated | 15 | 13

10. Secondary Outcome: Pre-dose Concentration of Afatinib in Plasma at Steady State on Day 29 (Cpre,ss,29)
Description: Cpre,ss,29 represents the pre-dose concentration of afatinib in plasma at steady state on day 29.
Time Frame: day 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 10 | 6
ng/mL | 33.1 (110) | 22.9 (64.7)

ADVERSE EVENTS:
Time Frame: First administration of trial medication until 28 days after last administration of trial medication
Arm/Group | Cohort A | Cohort B
Serious Adverse Events (participants affected / at risk) | 13/29 | 7/21
Other Adverse Events (participants affected / at risk) | 28/29 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=29) | Cohort B (N=21)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 1 | 0
Eyelid ptosis (Eye disorders) | 1 | 0
Miosis (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 5 | 0
Mucosal inflammation (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Abscess rupture (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
VIth nerve paralysis (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=29) | Cohort B (N=21)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0
Blepharitis (Eye disorders) | 0 | 2
Conjunctivitis (Eye disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 25 | 16
Dysphagia (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 13 | 5
Oral pain (Gastrointestinal disorders) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 5 | 2
Vomiting (Gastrointestinal disorders) | 4 | 6
Fatigue (General disorders) | 9 | 7
Mucosal inflammation (General disorders) | 9 | 6
Pain (General disorders) | 1 | 2
Weight decreased (Investigations) | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 8 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Dysgeusia (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 11 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 4
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 9 | 10
Skin fissures (Skin and subcutaneous tissue disorders) | 2 | 3
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication